CLINICAL TRIAL: NCT04030273
Title: Prevalence of Intrauterine Adhesions After Abdominal Myomectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: ADAM-1
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Myoma;Uterus
Keywords: Intrauterine adhesions; Abdominal myomectomy; Hysteroscopy
MeSH Terms: conditions — Myofibroma; Gynatresia | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open (laparotomic) myomectomy: Women undergoing uterine myomectomy by open surgery (laparotomy).
  Interventions: Diagnostic Test: Diagnostic hysteroscopy
- Laparoscopic myomectomy: Women undergoing uterine myomectomy by laparoscopy.
  Interventions: Diagnostic Test: Diagnostic hysteroscopy
- Robotic myomectomy: Women undergoing uterine myomectomy by robotic surgery.
  Interventions: Diagnostic Test: Diagnostic hysteroscopy

INTERVENTIONS:
Diagnostic Test: Diagnostic hysteroscopy — Diagnostic hysteroscopy performed in outpatient setting, using "no touch" vaginoscopy technique with a 2.9 mm 30-degree rigid hysteroscope with a single inflow sheet using normal saline as distention media.

SUMMARY:
Uterine fibroids are the most common benign tumors of the genital organs of women of childbearing age. Literature data show that more than 75% of women have fibroids.Symptomatic fibroids account for approximately over 200,000 hysterectomies and 50,000 myomectomies annually in the United States. Fibroids have a major impact on fertility, with significant adverse effect on implantation rate and spontaneous abortion rates when compared with infertile women without fibroids. The definitive treatment for uterine fibroids in a fertile patient is surgical excision. Although usually effective, myomectomy is not a risk-free operation, since the surgical procedure can cause mechanical infertility and can be associated with infection, injury to adjacent tissues, hemorrhage and need to convert to hysterectomy. A not often mentioned consequence of myomectomy is post-operative intrauterine adhesion formation. It has been reported that 50% of women undergoing open myomectomy are found to have intrauterine adhesions diagnosed by hysteroscopy performed 3 months after surgery. Such a high prevalence of intrauterine adhesions after open myomectomy is unexpected, however only few studies have addressed this topic.

It is accepted that injury to the endometrium is generally considered to be the primary causative factor for the development of intrauterine adhesions. The reason for such a high incidence of intrauterine adhesions after open myomectomy is unclear. It is speculated that infection or in adverted closure of the uterine cavity may play a role in intrauterine adhesion formation. The relationship between the number of fibroids removed and the risk of adhesions suggests a traumatic etiology. In the preservation of the uterus for the purpose of fertility, it is essential to also understand the impact of myomectomy on the endometrium. Currently no guideline recommends in office hysteroscopy as follow-up after myomectomy. The purpose of the present study is to evaluate the frequency of uterine adhesions following myomectomy and the impact of number, size and location of the fibroids as well as intraoperative breach of the endometrial cavity at the time of the myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one or more uterine myomas
* Desire to preserve fertility/uterus
* Myomectomy (by laparotomy, laparoscopy or robotic approach).

Exclusion Criteria:

* Adults unable to consent
* Pregnant women
* Prisoners
* History of previous intrauterine procedures such as dilation and curettage
* History of known intrauterine adhesions
* History of documented pelvic inflammatory disease
* History of endometritis (acute or chronic)
* Hysteroscopic myomectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients from 18 to 45 years of age with the diagnosis of uterine fibroids, wish to preserve fertility/uterus, not candidates for hysteroscopic myomectomy who are scheduled to undergo laparoscopic, robotic assisted or open myomectomy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Intrauterine adhesions | 3 months after myomectomy
  Presence of intrauterine adhesion, following the American Fertility Society classification (Fertil Steril. 1988;49:944-955.) in mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carugno, Study Director — University of Miami; Andrea Tinelli, Study Chair — Vito Fazzi Hospital; Antonio Simone Laganà, Study Chair — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lagana AS, Garzon S, Dababou S, Uccella S, Medvediev M, Pokrovenko D, Babunashvili EL, Buyanova SN, Schukina NA, Shcherbatykh Kaschchuk MG, Kosmas I, Licchelli M, Panese G, Tinelli A. Prevalence of Intrauterine Adhesions after Myomectomy: A Prospective Multicenter Observational Study. Gynecol Obstet Invest. 2022;87(1):62-69. doi: 10.1159/000522583. Epub 2022 Feb 15. PMID 35168241